CLINICAL TRIAL: NCT02039895
Title: Helical Irradiation of Total Skin (HITS) for Cutaneous Lymphoma
Acronym: HITS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FEMH-IRB-102135-F
Record Dates: First submitted 2014-01-15; First posted 2014-01-20 (Estimated); Last update posted 2014-08-04 (Estimated); Status verified 2014-01

CONDITIONS: Cutaneous T-cell Lymphoma
Keywords: Cutaneous T-cell lymphoma; Helical irradiation of the total skin; Refractory; Total skin electron beam therapy
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HITS for CTCL (Experimental): Cutaneous T-cell lymphoma treats by helical irradiation of the total skin (HITS) using helical tomotherapy
  Interventions: Radiation: HITS

INTERVENTIONS:
Radiation: HITS — Helical irradiation of the total skin by helical tomotherapy

SUMMARY:
Radiation therapy, Total skin electron beam therapy (TSEBT), achieves a high response rate and is an effective treatment for cutaneous T-cell lymphoma affecting the superficial region. One the most widely used TSEBT techniques consists of six dual fields initially developed at Stanford University. However, deviations occur from the prescription dose up to 40% and the surface dose inhomogeneity as much as 90% in body areas such as the perineum and eyelid.

Helical tomotherapy (HT) has advantages in irradiating extended volumes with treatment length of up to 160 cm, continuously in a helical pattern without the need for field junction. Using HT, an image-guided intensity-modulated radiotherapy, to replace conventional TSEBT technique to increase dose delivery and decrease toxicities possibly. Recently, we published the possibility of helical irradiation of the total skin (HITS) by physical proving and showed the clinical results of HITS successfully for a woman with T cell lymphoma failure by chemotherapy, topic UV irradiation and local radiotherapy (RT) to overcome the surface dose inhomogeneity by conventional RT.

Here, investigators will enroll the stage I-IV cutaneous T-cell lymphoma (CTCL) of International Society Cutaneous Lymphomas (ISCL)/U.S. Cutaneous Lymphoma Consortium (USCLC)/European Organization for Research & Treatment of Cancer (EORTC), patients who are candidates for TSEBT by recommendation of National Comprehensive Cancer Network Guidelines (Version 4.2011, Mycosis fungoid/Sezary syndrome) or who are refractory or not feasible to the topic UV irradiation, Interferon alpha, psoralen plus ultraviolet A photochemotherapy, and Accutane® (Isotretinoin) or chemotherapy to receive HITS to replace TSEBT. Additionally, we will compare the advantages and disadvantages between the plan of HT and conventional RT for TSEBT.

ELIGIBILITY:
Inclusion Criteria:

1. The stage I-IV cutaneous T-cell lymphoma (CTCL) of International Society Cutaneous Lymphomas (ISCL) and U.S. Cutaneous Lymphoma Consortium (USCLC)/European Organization for Research & Treatment of Cancer (EORTC), patients who are candidates for TSEB by recommendation of National Comprehensive Cancer Network Guidelines (Version 4.2011, Mycosis fungoid/Sezary syndrome)
2. Patients who are refractory or not feasible to the topic UV irradiation, Interferon alpha, psoralen plus ultraviolet A photochemotherapy, and Isotretinoin or chemotherapy.
3. Eligibility criteria included the following: Karnofsky status 70% or greater; creatinine clearance greater than 50 mL/min; cardiac left ventricular ejection fraction 50% or greater; aspartate aminotransferase and alanine aminotransferase less than 2.5 times the upper limits of institutional normal; adequate pulmonary function as shown by a forced expiratory volume of greater than 60%; and peripheral neuropathy grade 1 or lower. Patients were preassessed for their ability to lie supine for approximately 1 hour.
4. They had to be previously untreated TSEBT. Prior local radiation was permitted.
5. All patients voluntarily signed an informed consent form approved by the Institutional Review Board.

Exclusion Criteria:

1. Patient were prior treated by TSEBT for CTCL, another type of cancer, abnormal cardiac function (systolic ejection fraction < 50 percent or an abnormal stress test), chronic respiratory disease (vital capacity or carbon monoxide diffusion, < 50 percent of normal), abnormal liver function (serum bilirubin, > 2.0 mg per deciliter [>35 micromol per liter]; or serum aminotransferase values more than four times the normal value), and psychiatric disease.
2. Females who are pregnant/lactating or planning to be pregnant.
3. Patients with other systemic diseases that required long-term (≥ 2 weeks) usage of glucocorticosteroid or immunosuppressant agent(s) within 4 weeks prior to the initiation of study treatment.
4. Child or handicap are excluded

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Serious and Non-Serious Adverse Events | 3 months
  participants will be followed from the duration of RT to RT finish 1 month, an expected average of 3 ms

SECONDARY OUTCOMES:
Time to Disease Progression | Up to 24 ms

CONTACTS AND LOCATIONS:
Overall Officials: Chen-Hsi Hsieh, M.D., Ph.D., Study Director — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Taiwan